CLINICAL TRIAL: NCT01778361
Title: HIV UPBEAT: Understanding the Pathology of Bone Disease in HIV-infected. A Prospective Cohort Study of HIV-infected Patients and HIV-negative Subjects.
Brief Title: HIV UPBEAT: Understanding the Pathology of Bone Disease in HIV-infected Patients.
Acronym: UPBEAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College Dublin (Other)
Collaborators: Health Research Board, Ireland (Other)
Responsible Party: Principal Investigator, Patrick Mallon, Associate Dean of Post-graduate Research, School of Medicine and Medical Sciences, Head of HIV Molecular Research Group, Consultant Infectious Diseases., University College Dublin
Other Study IDs: HIVUPBEAT
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Osteoporosis
Keywords: Human immunodeficiency virus; low bone mineral density; osteopenia; osteoporosis; fracture
MeSH Terms: conditions — Osteoporosis; Acquired Immunodeficiency Syndrome; Bone Diseases, Metabolic; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, buffy coat, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV positive
- HIV negative

SUMMARY:
Despite the prevalence of osteopenia and osteoporosis in the HIV positive population, relatively little is known about the underlying pathology. This prospective cohort study aims to gain further understanding about a number of issues relating to low bone mineral density in HIV-infected subjects.

DETAILED DESCRIPTION:
This study will follow HIV positive and negative subjects annually for 5 years. The aims of this study include:

* to describe the pathology underlying low bone mineral density
* to assess the relationship between low bone mineral density and antiretroviral therapy exposure
* to assess the relationship between low bone mineral density and vitamin D /PTH status and/or markers of bone metabolism
* to assess the relationship between osteopenia and subsequent changes in bone mineral density and markers of bone metabolism
* to assess the validity of the currently available fracture risk assessment tool in predicting fractures in HIV positive populations

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* be able to provide written, informed consent
* be able to attend the research centre in a fasting state and undergo DEXA scanning

Exclusion Criteria:

* Subjects on bisphosphonate therapy at screening
* Pregnant or breastfeeding female subjects
* Subjects with a previous clinical history of primary hyperthyroidism or HIV negative subjects with elevated parathyroid hormone at screening
* HIV-negative subjects with a prior history of osteoporosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV positive patients and HIV negative subjects
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-02; Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Bone pathology | 3 years
  To describe abnormalities in bone pathology in bone biopsies from HIV-infected subjects with low bone mineral density by comparing biopsy indices to reference ranges.

SECONDARY OUTCOMES:
Rates of change in bone mineral density | 3 years
  To determine rates of change in bone mineral density in HIV-positive patients compared to HIV-negative controls

OTHER OUTCOMES:
Fracture incidence | 3 years
  To assess the validity of currently available fracture risk assessment tools in predicting fracture risk in HIV-infected patients.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick WG Mallon, MB BCh, BSc, PhD, Principal Investigator — HIV Molecular Research Group, University College Dublin
Locations (1):
- Mater Misericordiae University Hospital, Dublin, Ireland